CLINICAL TRIAL: NCT03519815
Title: Prospective Randomized Study to Evaluate the Efficacy and Tolerability of Ectoin® Containing Eye Spray (EES09) and Comparison to the Liposomal Eye Spray Tears Again® (TA) in the Treatment of Dry Eye Disease
Brief Title: Clinical Study to Evaluate the Efficacy of Ectoin® Containing Eye Spray for Treatment of Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Responsible Party: Principal Investigator, Daniela Nosch, Prof. Dr., University of Applied Sciences and Arts Northwestern Switzerland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-00462
Record Dates: First submitted 2018-04-16; First posted 2018-05-09 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Dry Eye
Keywords: dry eye; eye spray
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ectoin Eye Spray (Active Comparator): Eye Spray to be applied 3 times per day for the duration of 10 +/-3 days "Ectoin® Eye Spray - Colloidal" (EES09; bitop AG) - CE marked medical device
  Ingredients: Ectoin®, Soy-Lecithin, Vitamin A, Vitamin E, water, physiological buffer system Indication: to treat mild to moderate dry eye disease
  Interventions: Device: Ectoin® Eye Spray - Colloidal
- Liponit Eye Spray (Active Comparator): Eye Spray to be applied 3 times per day for the duration of 10 +/-3 days
  Liposomal eye spray: Tears Again® (TA, Optima Medical Swiss AG) - CE marked medical device Ingredients: Soy-Lecithin, Sodium Chloride, Ethanol, Phenoxyethanol, Vitamin A-Palmitate, Vitamin E, Aqua purificata Indication: to treat mild to moderate dry eye disease
  Interventions: Device: Liposomal eye spray Tears Again®

INTERVENTIONS:
Device: Ectoin® Eye Spray - Colloidal — eye spray to be applied to the closed eye lid
  Arms: Ectoin Eye Spray
Device: Liposomal eye spray Tears Again® — eye spray to be applied to the closed eye lid
  Arms: Liponit Eye Spray

SUMMARY:
Subjective and objective evaluation of the efficacy and tolerability of preservative-free "Ectoin® Eye Spray - Colloidal" and comparison of the efficacy and tolerability between "Ectoin® Eye Spray - Colloidal" and Tears Again® in patients with mild-moderate dry eye disease

DETAILED DESCRIPTION:
"Dry eye is a multifactorial disease of the ocular surface characterized by a loss of homeostasis of the tear film, and accompanied by ocular symptoms, in which tear film instability and hyperosmolarity, ocular surface inflammation and damage, and neuro- sensory abnormalities play etiological roles." (DEWS II Report, 2017).

For the treatment and prevention of dry eye disease (DED) there are a number of treatment modalities available, depending on the severity and classification (aqueous deficient / evaporative) of the disease. The liposomal eye spray Tears Again® (TA, Optima Medical Swiss AG - medical device with CE marking) represents an option to treat mild to moderate evaporative DED. A novel preservative-free eye spray, Ectoin® Eye Spray - Colloidal (EES09; bitop AG -medical device with CE marking), was developed, in which colloids (colloidal lecithin emulsion) serve as a carrier for Ectoin. Ectoin is known as a natural cell-protective and inflammatory-inhibiting molecule. The principle mode of action of Ectoin is based on the physical interaction of this compatible solute with water and the resulting effects of the Ectoin-Hydro-Complex on the tissue treated.

The aim of this study is to subjectively and objectively evaluate the efficacy and tolerability of preservative-free "Ectoin® Eye Spray - Colloidal" and to compare the efficacy and tolerability between "Ectoin® Eye Spray - Colloidal" and Tears Again® in patients with mild-moderate dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years
* OSDI Score of at least 18
* NIBUT smaller or equal to 10s in at least one eye

Exclusion Criteria:

* Post-operative trauma or injury
* Ocular disease with exception of DED
* Hypersensitivity to any of the ingredients in the products used for this study
* Contact lens wear 24h before or on the day of study visits
* Use of eye drops / other eye sprays on the day of visit 1 or during the duration of the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in subjective variables 10min after application and after the treatment period with the eye sprays, in comparison to baseline measurements (visit 1). | 10min
  ocular surface disease index (OSDI) questionnaire, VAS questionnaire for evaluation of dry eye symptoms and tolerability of the eye spray.
Difference in tear film quality | 10min
  non-invasive tear film break up time (NIBUT)
Difference in tear film osmolarity | 10min
  osmolarity measurement
Difference in conjunctival bulbar redness | 10min
  grading of conjunctival bulbar redness

SECONDARY OUTCOMES:
Difference in subjective variables after the treatment period between the two eye sprays. | 10 +/- 3 days
  ocular surface disease index (OSDI) questionnaire, VAS questionnaire for evaluation of dry eye symptoms and tolerability of the eye spray.
Difference in tear film quality | 10 +/- 3 days
  non-invasive tear film break up time (NIBUT)
Difference in tear film osmolarity | 10 +/- 3 days
  osmolarity measurement
Difference in conjunctival bulbar redness | 10 +/- 3 days
  grading of conjunctival bulbar redness

CONTACTS AND LOCATIONS:
Overall Officials: Daniela S Nosch, PhD, Principal Investigator — University of Applied Sciences and Arts Northwestern Switzerland
Locations (1):
- Institute of Optometry, FHNW, Olten, Canton of Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig JP, Purslow C, Murphy PJ, Wolffsohn JS. Effect of a liposomal spray on the pre-ocular tear film. Cont Lens Anterior Eye. 2010 Apr;33(2):83-7. doi: 10.1016/j.clae.2009.12.007. Epub 2010 Jan 21. PMID 20096622
- [Result] Craig JP, Nelson JD, Azar DT, Belmonte C, Bron AJ, Chauhan SK, de Paiva CS, Gomes JAP, Hammitt KM, Jones L, Nichols JJ, Nichols KK, Novack GD, Stapleton FJ, Willcox MDP, Wolffsohn JS, Sullivan DA. TFOS DEWS II Report Executive Summary. Ocul Surf. 2017 Oct;15(4):802-812. doi: 10.1016/j.jtos.2017.08.003. Epub 2017 Aug 8. PMID 28797892
- [Result] Dausch D, Lee S, Dausch S, Kim JC, Schwert G, Michelson W. [Comparative study of treatment of the dry eye syndrome due to disturbances of the tear film lipid layer with lipid-containing tear substitutes]. Klin Monbl Augenheilkd. 2006 Dec;223(12):974-83. doi: 10.1055/s-2006-927266. German. PMID 17199193
- [Result] Lee S, Dausch S, Maierhofer G, Dausch D. [A new therapy concept for the treatment of dry eye--the usefulness of phospholipid liposomes]. Klin Monbl Augenheilkd. 2004 Oct;221(10):825-36. doi: 10.1055/s-2004-813715. German. PMID 15499517
- [Result] Khaireddin R, Schmidt KG. [Comparative investigation of treatments for evaporative dry eye]. Klin Monbl Augenheilkd. 2010 Feb;227(2):128-34. doi: 10.1055/s-0028-1109686. Epub 2009 Sep 15. German. PMID 19757354